CLINICAL TRIAL: NCT05894148
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-dose Escalation Phase I Study of Genakumab for Injection in Chinese Healthy Adults
Brief Title: Clinical Study of Multiple Dose Genakumab for Injection in Chinese Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Afﬁliated Hospital of North Sichuan Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GenSci048-102
Record Dates: First submitted 2023-02-27; First posted 2023-06-08 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Interstitial Lung Disease
Keywords: Safety,; Tolerability,; Pharmacokinetics,; Genakumab
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genakumab injection (Experimental): Group 1: 120mg，group 2: 200mg
  Interventions: Drug: Genakumab injection
- placebo (Placebo Comparator): The placebo contains other excipients except Genakumab, and its appearance is consistent with that of Genakumab for injection
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Genakumab injection — Group 1: 120mg Q4W，group 2: 200mg Q4W
  Arms: Genakumab injection
Drug: placebo — The placebo contains other excipients except Genakumab, and its appearance is consistent with that of Genakumab for injection.
  Arms: placebo

SUMMARY:
To evaluate the safety and tolerability of multiple-dose subcutaneous injections of Genakumab for Injection in Chinese healthy adult volunteers.

DETAILED DESCRIPTION:
There are 2 dose groups with 12 participants in each group, including 10 participants in the experimental group and 2 participants in the placebo control group. Each subject receives Genakumab or placebo once every four weeks for three times.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ age ≤45 years, and in good health;
* body mass index is within the range of 19 - 26 kg/m^2 (including 19 kg/m^2 and 26 kg/m^2);
* No parental scheme from the screening period to 3 months after the study period.

Exclusion Criteria:

* Participants have abnormal physical and auxiliary examination results with clinical significance;
* History of cardiovascular, liver, kidney, digestive, blood, nervous system and allergic diseases, mental and metabolic disorders,
* Participants who use any prescription drugs within 2 weeks prior dosing.
* Participants who receive (attenuated) live vaccines within 3 months prior to dosing;
* Participation in any clinical investigation within 3 months prior to dosing;
* Donation or loss of 400 mL or more of blood within 3 months prior to dosing;
* Tuberculosis symptoms, contact with patients with suspected tuberculosis symptoms
* Positive results in Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, Syphilis antibody or HIV antibody;
* Current or previous drug or alcohol abuse;
* Other conditions in which the investigator preclude enrollment into the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
The frequency of adverse events (AE) | Up to 20 weeks
  adverse events during the study are to assess the safety of Genakumab.

SECONDARY OUTCOMES:
Maximum observed serum Genakumab concentration | up to 20 weeks
  This is to assess pharma co kinetics of Genakumab.
Area under the serum Genakumab concentration-time curve | up to 20 weeks
  This is to assess pharma co kinetics of Genakumab.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolan Yong, bachelor, Study Chair — Chengdu Xinhua Hospital
Locations (1):
- Chengdu Xinhua Hospital Affiliated to North Sichuan Medical College, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No